CLINICAL TRIAL: NCT00048932
Title: A Phase III Study of BMS-188667 in Subjects With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-031
Record Dates: First submitted 2002-11-11; First posted 2002-11-13 (Estimated); Results first posted 2011-05-03 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Double-blind abatacept (Active Comparator): Participants received a fixed dose of abatacept approximating 10 mg/kg (500 mg for participants < 60 kg, 750 mg for participants 60 to 100 kg and 1 g for participants > 100 kg). Abatacept was administered intravenously (IV) on Days 1, 15, 29, and every 28 days thereafter, for a total of 14 doses. Participants also received background therapy(ies) for rheumatoid arthritis (RA) (non-biologic or biologic disease-modifying drugs [DMARDs], or combination) throughout the double-blind treatment period
  Interventions: Drug: Double-blind Abatacept
- Double-blind Placebo (Placebo Comparator): Participants received Placebo (dextrose 5% water [D5W] for injection U.S.P or normal saline [NS]) for IV infusion administered on Days 1, 15, 29, and every 28 days thereafter, for a total of 14 doses. Participants also received background therapy(ies) for rheumatoid arthritis (RA) (non-biologic or biologic disease-modifying drugs [DMARDs], or combination) throughout the double-blind treatment period.
  Interventions: Drug: Double-blind Placebo
- Open-label Abatacept (Active Comparator): Participants received abatacept (weight-tiered 10 mg/kg dose) IV every 28 days during the open-label period.
  Interventions: Drug: Open-label Abatacept

INTERVENTIONS:
Drug: Double-blind Abatacept — Concentrate and diluted in a solution, IV, 500 mg (body weight < 60 Kg); 750 mg (body weight 60-100 Kg); 1000 mg (body weight > 100 Kg), Once daily, Day 1, 15, and 29.
  Other Names: Orencia; BMS-188667
  Arms: Double-blind abatacept
Drug: Double-blind Placebo — Concentrate and diluted in a solution, IV, 0 mg, Once daily, Day 1, 15, and 29.
  Arms: Double-blind Placebo
Drug: Open-label Abatacept — Concentrate and diluted in a solution, IV, 500 mg (body weight < 60 Kg); 750 mg (body weight 60-100 Kg); 1000 mg (body weight > 100 Kg), Once daily, Every 28 days.
  Other Names: Orencia; BMS-188667
  Arms: Open-label Abatacept

SUMMARY:
The purpose of this clinical research study is to learn if abatacept is safe when co-administered with other approved rheumatoid arthritis medications.

DETAILED DESCRIPTION:
This was a multinational, multicenter, randomized, double-blind, 2-arm, parallel-dosing designed study. The treatment period was 12 months. Eligible participants were randomized to 1 of 2 treatment groups: abatacept fixed dose approximating 10 mg/kg (based on participant's body weight; 500 mg for participants weighing < 60kg; 750 mg for participants weighing 60 to 100 kg; and 1 gram for participants weighing > 100 kg, monthly) or placebo intravenous (IV) infusion. All participants continued their background therapy(ies) for rheumatoid arthritis (RA) (non-biologic or biologic disease-modifying drugs [DMARDs], or combination) throughout the double-blind treatment period. Double-blind study medication (abatacept or placebo) was administered on Days 1, 15, 29, and every 28 days thereafter, for a total of 14 doses.

All participants who completed the 12-month double-blind study period (Day 1 through Day 365), were eligible to continue into the open-label period. All eligible participants (active or placebo) were re-allocated to receive abatacept at a weight-tiered dose that approximated 10 mg/kg, based on their Day 365 body weight. Participants continued to receive infusions every 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria of American Rheumatism Association for the diagnosis of rheumatoid arthritis and the American College of Rheumatology functional classes I, II III or IV
* Participants must be taking 1 or more DMARDs and/or biologic approved for rheumatoid arthritis (RA) for at least 3 months and be on a stable dose for 28 days prior to Day 1.

Exclusion:

* Other auto-immune disease as a main diagnosis (e.g. Systemic Lupus Erythematosus [SLE], Scleroderma)
* Active tuberculosis (TB) requiring treatment within last 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1795 (Actual)
Dates: Start 2002-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Local Institution, Decatur, Alabama
  - Local Institution, Paradise, Arizona
  - Local Institution, Phoenix, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, San Francisco, California
  - Local Institution, Loveland, Colorado
  - Local Institution, Hamden, Connecticut
  - Local Institution, Lake Worth, Florida
  - Local Institution, Largo, Florida
  - Local Institution, Blairsville, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Evansville, Indiana
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Wichita, Kansas
  - Local Institution, Louisville, Kentucky
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Baltimore, Maryland
  - Local Institution, Cumberland, Maryland
  - Local Institution, Westminster, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, Grand Rapids, Michigan
  - Local Institution, Royal Oak, Michigan
  - Local Institution, Toms River, New Jersey
  - Local Institution, Los Alamos, New Mexico
  - Local Institution, New York, New York
  - Local Institution, Durham, North Carolina
  - Local Institution, Hickory, North Carolina
  - Local Institution, Canton, Ohio
  - Local Institution, Cleveland, Ohio
  - Local Institution, Columbus, Ohio
  - Local Institution, Elyria, Ohio
  - Local Institution, Youngstown, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Wyomissing, Pennsylvania
  - Local Institution, Columbia, South Carolina
  - Local Institution, Sioux Falls, South Dakota
  - Local Institution, Ducktown, Tennessee
  - Local Institution, Nashville, Tennessee
  - Local Institution, Richmond, Virginia
  - Local Institution, Edmonds, Washington
  - Local Institution, Olympia, Washington
  - Local Institution, Tacoma, Washington
  - Local Institution, Menomonee Falls, Wisconsin
  - Local Institution, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Alten R, Burkhardt H, Feist E, Kruger K, Rech J, Rubbert-Roth A, Voll RE, Elbez Y, Rauch C. Abatacept used in combination with non-methotrexate disease-modifying antirheumatic drugs: a descriptive analysis of data from interventional trials and the real-world setting. Arthritis Res Ther. 2018 Jan 2;20(1):1. doi: 10.1186/s13075-017-1488-5. PMID 29329602

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1795 enrolled in study and 339 were not randomized due to no longer meeting study criteria (n=214), withdraw of consent (n=83), other reasons (n=32), participant was lost to follow-up (n=5), administrative reason by sponsor (n=2), adverse event (n=2), and poor/non-compliance (n=1). Of 1456 randomized, 15 were not treated.
Groups:
- Abatacept (ABA): Participants received a fixed dose of abatacept approximating 10 mg/kg (500 mg for participants < 60 kg, 750 mg for participants 60 to 100 kg and 1 g for participants > 100 kg). Abatacept was administered intravenously (IV) on Days 1, 15, 29, and every 28 days thereafter, for a total of 14 doses. Participants also received background therapy(ies) for rheumatoid arthritis (RA) (non-biologic or biologic disease-modifying drugs [DMARDs], or combination) throughout the double-blind treatment period.
- Placebo (PLA): Participants received Placebo (dextrose 5% water [D5W] for injection U.S.P or normal saline [NS]) for IV infusion administered on Days 1, 15, 29, and every 28 days thereafter, for a total of 14 doses. Participants also received background therapy(ies) for rheumatoid arthritis (RA) (non-biologic or biologic disease-modifying drugs [DMARDs], or combination) throughout the double-blind treatment period.
- Open Label (OL) Abatacept: Participants received abatacept (weight-tiered 10 mg/kg dose) IV every 28 days during the open-label period.
Period: Double Blind Period (DB)
Arm/Group | Abatacept (ABA) | Placebo (PLA) | Open Label (OL) Abatacept
Started | 959 (Number Treated) | 482 (Number Treated) | 0
Completed | 836 | 395 | 0
Not Completed | 123 | 87 | 0
Not completed — Administrative Reason By Sponsor | 1 | 0 | 0
Not completed — Adverse Event | 51 | 19 | 0
Not completed — Death | 5 | 3 | 0
Not completed — Lack of Efficacy | 26 | 44 | 0
Not completed — Lost to Follow-up | 3 | 4 | 0
Not completed — Relocation | 1 | 0 | 0
Not completed — Uncontrolled hypertension | 0 | 1 | 0
Not completed — Missed 2 doses while undergoing work-up | 1 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — No Longer Meets Study Criteria | 8 | 2 | 0
Not completed — Withdrawal by Subject | 24 | 10 | 0
Not completed — Poor/Non-Compliance | 2 | 4 | 0
Period: Open Label Period (OL)
Arm/Group | Abatacept (ABA) | Placebo (PLA) | Open Label (OL) Abatacept
Started | 0 | 0 | 1184 (47 participants who completed the double-blind did not enter the open-label)
Completed | 0 | 0 | 743
Not Completed | 0 | 0 | 441
Not completed — Death | 0 | 0 | 25
Not completed — Adverse Event | 0 | 0 | 103
Not completed — Lack of Efficacy | 0 | 0 | 81
Not completed — Lost to Follow-up | 0 | 0 | 27
Not completed — Withdrawal by Subject | 0 | 0 | 117
Not completed — No Longer Meets Study Criteria | 0 | 0 | 5
Not completed — Poor/Non-Compliance | 0 | 0 | 13
Not completed — Pregnancy | 0 | 0 | 6
Not completed — Administrative Reason By Sponsor | 0 | 0 | 20
Not completed — Investigator Retiring | 0 | 0 | 2
Not completed — Participant Transportation Issues | 0 | 0 | 1
Not completed — Participant Relocated | 0 | 0 | 6
Not completed — Investigator Dosing the Trial | 0 | 0 | 1
Not completed — Site Closure | 0 | 0 | 3
Not completed — Trial Terminated | 0 | 0 | 1
Not completed — Difficult IV Access with Participant | 0 | 0 | 1
Not completed — Patient Decision | 0 | 0 | 4
Not completed — Participant Received Wrong Medication | 0 | 0 | 1
Not completed — Participant Desires Pregnancy | 0 | 0 | 2
Not completed — Participant Missed Consecutive Doses | 0 | 0 | 5
Not completed — Medication Lost Efficacy | 0 | 0 | 1
Not completed — Investigator Decision | 0 | 0 | 4
Not completed — Site Staff Issues | 0 | 0 | 2
Not completed — Site Not Participating in Open Label | 0 | 0 | 9
Not completed — Participant Surgery | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept (ABA) | Placebo (PLA) | Total
Number analyzed (Participants) | 959 | 482 | 1441
Age Continuous [Mean (Standard Deviation); unit: years] | 52.4 (11.7) | 52.1 (12.0) | 52.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 789 | 398 | 1187
  Male | 170 | 84 | 254

OUTCOME MEASURES:

1. Primary Outcome: Double Blind Period (DB); Number of Participants With Death, Serious Adverse Events (SAEs), Related SAEs, SAEs Leading to Discontinuation, Adverse Events (AEs), Related AEs, or AEs Leading to Discontinuation
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event. Related SAE/AE = possibly, probably, or certainly related to study drug
Time Frame: Day 1 to Day 365, and including data up to 56 days post last dose of double-blind medication
Population: All Treated Participants, all participants who received at least 1 dose of study medication
Measure: Number; unit: participants
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 959 | 482
participants
  Death | 5 | 4
  SAEs | 123 | 59
  Related SAEs | 23 | 13
  SAEs Leading to Discontinuation | 23 | 7
  AEs | 866 | 417
  Related AEs | 534 | 239
  AEs Leading to Discontinuation | 52 | 20

2. Primary Outcome: DB; Number of Participants With AEs of Special Interest
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. AEs of special interest are those AEs that may be associated with the use of immunomodulatory drugs, including all infections, serious infections, and opportunistic infections; autoimmune disorders; neoplasms; acute infusional AEs (pre-specified AEs occurring within 1 hour of start of infusion) and peri-infusional AEs (pre-specified AEs occurring within 24 hours of the start of infusion).
Time Frame: Day 1 to Day 365, and including data up to 56 days post last dose of double-blind medication
Population: All Treated Participants, all participants who received at least 1 dose of study medication
Measure: Number; unit: participants
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 959 | 482
participants
  Infections/Infestations | 95 | 40
  Serious Infections/Infestations | 17 | 5
  Neoplasms | 34 | 17
  Pre-specified Autoimmune Disorders | 32 | 15
  Pre-specified Acute Infusional AEs | 96 | 34
  Pre-specified Peri-Infusional AEs | 233 | 98

3. Primary Outcome: DB; Number of Participants With Hematology Laboratories Meeting Marked Abnormality Criteria
Description: Upper Normal Limit (ULN), Lower Normal Limit (LLN), Baseline (BL). Marked abnormality criteria are: Hemoglobin (HGB): >3 g/dL decrease from BL; Hematocrit: <0.75 * BL; Erythrocytes: <0.75 * BL; Platelets (PLT): <0.67 * LLN/>1.5 * ULN, or if BL < LLN then use <0.5 * BL and <100,000 mm^3; Leukocytes: <0.75 * LLN/ >1.25 * ULN, or if BL<LLN then use <0.8 * BL or >ULN, or if BL>ULN then use >1.2 * BL or <LLN; neutrophils+bands: <1.0 * 10^3 c/uL; eosinophils: >0.750 * 10^3 c/uL; basophils: > 400 mm^3; monocytes: >2000 mm^3; lymphocytes: <0.750 * 10^3 c/uL/ >7.50 * 10^3 c/uL.
Time Frame: Day 1 to Day 365, and including data up to 56 days post last dose of double-blind medication
Population: All Treated Population. One participant in each group was not evaluated for hematology abnormalities due to data unavailability (missing data).
Measure: Number; unit: participants
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 958 | 481
participants
  Low HGB (LLN=1.5%) | 12 | 14
  Low hematocrit (LLN=36%) | 9 | 12
  Low erythrocytes (LLN=3.72-4.27 x10*6 c/uL) | 0 | 0
  Low PLT (LLN=140-157*10^9 c/L) | 7 | 3
  High PLT (ULN=415-440*10^9 c/L) | 2 | 4
  Low leukocytes (LLN= 4-9*10^3 c/uL) | 24 | 12
  High leukocytes (ULN = 10.5-30*10^3 c/uL) | 70 | 57
  Low neutrophils + bands (LLN= 1.5-2.9*10^3 c/uL) | 16 | 9
  Low lymphocytes (LLN= 0.7-2.9*10^3 c/uL) | 0 | 0
  High lymphocytes (ULN= 4.5-13.3*10^3 c/uL) | 0 | 0
  High monocytes (ULN=1-3.9*10^3 c/uL) | 0 | 0
  High basophils (ULN= 0.6*10^3 c/uL) | 0 | 0
  High eosinophils (ULN= 1.5*10^3 c/uL) | 0 | 0

4. Primary Outcome: DB; Number of Participants With Blood Chemistry Laboratories Meeting Marked Abnormality (MA) Criteria
Description: ULN=upper level of normal; BL=baseline.Marked abnormality criteria: High alkaline phosphatase (ALP): >2* ULN, or if BL>ULN then use >3* BL; high aspartate aminotransferase (AST): >3* ULN (80 U/L), or if BL>ULN then use >4* BL; high alanine aminotransferase (ALT): >3* ULN (34-47 U/L), or if BL>ULN then use >4* BL; high G-Glutamyl transferase (GGT): >2* ULN, or if BL>ULN then use >3* BL; high bilirubin: >2* ULN, or if BL>ULN then use >4* BL; high blood urea nitrogen (BUN): >2* BL; high creatinine: >1.5* BL (ULN 14.6 pg/mg. AST ULN=80 U/L; ALT ULN=34-47 U/L;creatinine ULN=14.6 pg/mg.
Time Frame: Day 1 to Day 365, and including data up to 56 days post last dose of double-blind medication
Population: All Treated Population. Two participants in the ABA group and 3 participants in the PLA group were not evaluated for blood chemistry abnormalities due to data unavailability (missing data).
Measure: Number; unit: participants
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 957 | 479
participants
  High AST (ULN=80 U/L) | 12 | 3
  High ALT (ULN=34-47 U/L) | 16 | 9
  High creatinine (ULN=14.6 pg/mg) | 41 | 29

5. Secondary Outcome: DB; Number of Participants With Positive Anti-Abatacept or Anti-Cytotoxic T-Lymphocyte Antigen 4 (CTLA4) Responses by Enzyme-Linked Immunosorbant Assay (ELISA)
Description: Serum samples from all treated adult participants with active rheumatoid arthritis (RA) were screened for the presence of drug-specific antibodies using ELISA. Immunogenicity was defined as the presence of a positive anti-abatacept or anti-CTLA4 antibody.
Time Frame: Days 1, 29, 57, 85, 113,169, 281, 365
Population: All participants treated during DB who received at least 1 dose of abatacept and had antibody samples collected at baseline and at least 1 post-baseline visit. 561 participants were not evaluated for anti-abatacept anti-bodies during the DB.
Measure: Number; unit: participants
Groups:
- All Treated Participants: Participants received abatacept (weight-tiered 10 mg/kg dose) IV every 28 days during the open-label period.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 880
participants
  Anti-abatacept antibodies | 13
  Anti-CTLA4 antibodies | 9
  Total antibodies | 22

6. Primary Outcome: DB; Number of Participants With Clinically Significant Physical Examination or Vital Signs Abnormalities
Description: Physical examinations were performed at the discretion of the investigator and included breast examinations for female participants. Vital sign measurements were performed for participants before and after infusion of study medication at each visit and included seated systolic blood pressure, seated diastolic blood pressure, temperature, and heart rate. Abnormalities were determined to be clinically significant by the investigator.
Time Frame: Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, 337. Vital signs were measured at these visits before and after study medication infusion.
Population: All Treated Population.
Measure: Number; unit: participants
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 959 | 482
participants | 0 | 0

7. Primary Outcome: Open Label Period (OL); Number of Participants With Death, Serious Adverse Events (SAEs), Related SAEs, SAEs Leading to Discontinuation, Adverse Events (AEs), Related AEs, or AEs Leading to Discontinuation
Description: as for outcome 1
Time Frame: Day 365 to Day 1,821
Population: All Treated Participants
Measure: Number; unit: participants
Groups:
- OL ABA: Participants received abatacept (weight-tiered 10 mg/kg dose) IV every 28 days during the open-label period.
Arm/Group | OL ABA
Number analyzed (Participants) | 1184
participants
  Death | 32
  SAEs | 425
  Related SAEs | 124
  SAEs Leading to Discontinuation | 70
  AEs | 1123
  Related AEs | 737
  AEs Leading to Discontinuation | 103

8. Primary Outcome: OL; Number of Participants With AEs of Special Interest
Description: as for outcome 2
Time Frame: Day 365 to Day 1821
Population: All Treated Participants, all participants who received at least 1 dose of study medication
Measure: Number; unit: participants
Arm/Group | OL ABA
Number analyzed (Participants) | 1184
participants
  Infections/Infestations | 957
  Total Neoplasms | 168
  Malignant Neoplasms | 56
  Benign and Unspecified Neoplasms | 112
  Pre-specified Autoimmune Disorders | 67
  Pre-specified Acute Infusional AEs | 82
  Pre-specified Peri-Infusional AEs | 219

9. Primary Outcome: OL; Number of Participants With Hematology Laboratories Meeting Marked Abnormality Criteria
Description: as for outcome 3
Time Frame: Day 365 to Day 1821, and including data up to 56 days post last dose of double-blind medication
Population: All Treated Population.
Measure: Number; unit: participants
Arm/Group | OL ABA
Number analyzed (Participants) | 1184
participants
  Low HGB (LLN=1.5%) | 70
  Low hematocrit (LLN=36%) | 53
  Erythrocytes (LLN=3.72-4.27 x10*6 c/uL) | 25
  Low PLT (LLN=140-157*10^9 c/L) | 23
  High PLT (ULN=415-440*10^9 c/L) | 10
  Low leukocytes (LLN= 4-9*10^3 c/uL) | 110
  High leukocytes (ULN = 10.5-30*10^3 c/uL) | 162
  Low neutrophils + bands (LLN= 1.5-2.9*10^3 c/uL) | 31
  Low lymphocytes (LLN= 0.7-2.9*10^3 c/uL) | 220
  High lymphocytes (ULN= 4.5-13.3*10^3 c/uL) | 5
  High monocytes (ULN=1-3.9*10^3 c/uL) | 11
  High basophils (ULN= 0.6*10^3 c/uL) | 4
  High eosinophils (ULN= 1.5*10^3 c/uL) | 151

10. Primary Outcome: OL; Number of Participants With Liver Function Laboratories Meeting Marked Abnormality Criteria
Description: Marked abnormality criteria: Alkaline phosphatase (ALP): >2* ULN, or if BL>ULN then use >3* BL; aspartate aminotransferase (AST): >3* ULN, or if BL>ULN then use >4* BL; alanine aminotransferase (ALT): >3* ULN, or if BL>ULN then use >4* BL; G-Glutamyl transferase (GGT): >2* ULN, or if BL>ULN then use >3* BL; Bilirubin: >2* ULN, or if BL>ULN then use >4* BL; blood urea nitrogen (BUN): >2* BL; creatinine: >1.5* BL
Time Frame: Day 365 to Day 1821, and including data up to 56 days post last dose of double-blind medication
Population: All Treated Population. One participant was not evaluated for liver function abnormalities.
Measure: Number; unit: participants
Arm/Group | OL ABA
Number analyzed (Participants) | 1183
participants
  High ALP (ULN=150 U/L) | 12
  High AST (ULN=80 U/L) | 38
  High ALT (ULN=34-47 U/L) | 54
  High GGT (ULN=43-54 U/L) | 91
  High bilirubin (ULN=0.3 mg/dL) | 9
  High BUN (normal=4-25 mg/dL) | 108
  High creatinine (ULN=14.6 pg/mg) | 204

11. Primary Outcome: OL; Number of Participants With Electrolyte Laboratories Meeting Marked Abnormality Criteria
Description: Marked abnormality criteria: Sodium (Na): <0.95*LLN/ >1.05*ULN, or if BL<LLN then use <0.95* BL or >ULN, or if BL>ULN then use>1.05* BL or <LLN; potassium (K): <0.9* LLN/>1.1*ULN, or if BL<LLN then use <0.9* BL or >ULN, or if BL>ULN then use>1.1* BL or <LLN; (Cl): <0.9* LLN/>1.1* ULN, or if BL<LLN then use <0.9* BL or >ULN, or if BL>ULN then use>1.1* BL or <LLN; calcium (Ca): <0.8* LLN/>1.2* ULN, or if BL<LLN then use <0.75* BL or >ULN, or if BL>ULN then use>1.25* BL or <LLN; phosphorous (P): <0.75* LLN/ >1.25* ULN, or if BL<LLN then use 0.67* BL or >ULN, or if BL>ULN then use>1.33* BL or <LLN
Time Frame: Day 365 to Day 1821, and including data up to 56 days post last dose of double-blind medication
Population: All Treated Population. One participant was not evaluated for electrolyte abnormalities.
Measure: Number; unit: participants
Arm/Group | OL ABA
Number analyzed (Participants) | 1183
participants
  Low Na (LLN=135 mEq/L) | 16
  High Na (ULN=148 mEq/L) | 1
  Low K (LLN=3.5 mEq/L) | 77
  High K (ULN=5.5 mEq/L) | 72
  Low Cl (LLN= 96 mEq/L) | 5
  High Cl (ULN=109 mEq/L) | 2
  Low Ca (LLN=8.5 mg/dL) | 2
  High Ca (ULN=11 mg/dL) | 0
  Low P (LLN=2.5 mg/dL) | 17
  High P (ULN 7.1 mg/dL) | 27

12. Primary Outcome: OL; Number of Participants With Other Chemistry and Urinalysis Laboratories Meeting Marked Abnormality Criteria
Description: MA criteria: serum glucose (Glu): <65 mg/dL/>220 mg/dL;fasting serum Glu: <0.8* LLN/>1.5*ULN,or if BL<LLN then use 0.8*BL or >ULN,or if BL>ULN then use >2.0*BL or <LLN;total protein: <0.9*LLN/>1.1*ULN,or if BL<LLN then use <0.9*BL or >UNL,or if BL>UNL then use >1.1*BL or <LLN; albumin: <0.9*LLN,or if BL<LLN then use <0.75 BL;uric acid: >1.5*ULN,or if BL>ULN then use >2*BL. Urinalysis (Urine protein,urine Glu,urine blood,leukocyte esterase,Red Blood Cells [RBCs], White Blood Cells [WBCs]):Use ≥2 when BL value missing or when pre-dose=0 or 0.5; use ≥3 when pre-dose=1, use ≥4 when pre-dose=2 or 3
Time Frame: Day 365 to Day 1821, and including data up to 56 days post last dose of double-blind medication
Population: All Treated Population. N=Number of Participants Analyzed, n=number of participants with measurements at time point
Measure: Number; unit: participants
Arm/Group | OL ABA
Number analyzed (Participants) | 1184
participants
  Low Glu, n=1184 | 207
  High Glu, n=1184 | 61
  Low fasting Glu, n=647 (LLN=65 mg/dL) | 647
  High fasting Glu, n=647 (ULN=115 mg/dL) | 41
  Low protein, n=1183 (LLN=6 g/dL) | 12
  High protein, n=1183 (ULN=8.5 g/dL) | 2
  Low albumin, n=1183 (LLN=3.5 g/dL) | 40
  High uric acid, n=1183 (ULN=8.7 mg/dL) | 19
  High urine protein, n=1184 (normal=trace) | 125
  High urine glucose, n=1184 (normal=negative) | 51
  High urine ketones, n=33 (normal=negative) | 0
  High urine blood, n=1184 (normal=negative) | 310
  High leukocyte esterase, n=32 | 12
  High urine WBC, n=852 | 429
  High urine RBC, n=852 | 403

13. Primary Outcome: OL; Number of Participants With Clinically Significant Physical Examination or Vital Signs Abnormalities
Description: as for outcome 6
Time Frame: Days 365 to Day 1821
Population: All Treated Population.
Measure: Number; unit: participants
Arm/Group | OL ABA
Number analyzed (Participants) | 1184
participants | 0

14. Secondary Outcome: DB; Number of Participants With Positive Anti-Abatacept or Anti-Cytotoxic T-Lymphocyte Antigen 4 (CTLA4) Responses by ELISA
Description: Serum samples from all treated adult participants with active rheumatoid arthritis were screened for the presence of drug-specific antibodies using ELISA. Immunogenicity was defined as the presence of a positive anti-abatacept or anti-CTLA4 antibody.
Time Frame: Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, 337
Population: All DB participants treated on study who received at least 1 dose of abatacept and had antibody samples collected at baseline and at least 1 post-baseline visit. 68 participants were not evaluated for anti-abatacept anti-bodies on study.
Measure: Number; unit: participants
Arm/Group | All Treated Participants
Number analyzed (Participants) | 1296
participants
  Anti-abatacept antibodies (n=1228) | 66
  Anti-CTLA4 antibodies (n=1296) | 48
  Total antibodies (n=1296) | 107

ADVERSE EVENTS:
Groups:
- Abatacept (ABA): Participants received a fixed dose of abatacept approximating 10 mg/kg (500 mg for subjects < 60 kg, 750 mg for subjects 60 to 100 kg and 1 g for subjects > 100 kg). Abatacept was administered intravenously (IV) on Days 1, 15, 29, and every 28 days thereafter, for a total of 14 doses. Participants also received background therapy(ies) for rheumatoid arthritis (RA) (non-biologic or biologic disease-modifying drugs [DMARDs], or combination) throughout the double-blind treatment period.
Arm/Group | Open Label (OL) Abatacept | Abatacept (ABA) | Placebo (PLA)
Serious Adverse Events (participants affected / at risk) | 425/1184 | 124/959 | 59/482
Other Adverse Events (participants affected / at risk) | 1010/1184 | 715/959 | 346/482
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label (OL) Abatacept (N=1184) | Abatacept (ABA) (N=959) | Placebo (PLA) (N=482)
CATARACT (Eye disorders) | 1 | 1 | 2
PTERYGIUM (Eye disorders) | 1 | 0 | 0
SCLEROMALACIA (Eye disorders) | 0 | 1 | 0
HIV TEST POSITIVE (Investigations) | 0 | 0 | 1
HAEMATOCRIT DECREASED (Investigations) | 1 | 0 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 0 | 0
TRANSAMINASES INCREASED (Investigations) | 1 | 0 | 0
ELECTROCARDIOGRAM CHANGE (Investigations) | 1 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0 | 0
ELECTROCARDIOGRAM ST-T SEGMENT ABNORMAL (Investigations) | 1 | 0 | 0
ARRHYTHMIA (Cardiac disorders) | 1 | 0 | 0
BRADYCARDIA (Cardiac disorders) | 0 | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1
PERICARDITIS (Cardiac disorders) | 1 | 0 | 0
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 3 | 2 | 1
CARDIOMYOPATHY (Cardiac disorders) | 1 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 3 | 0 | 0
ANGINA UNSTABLE (Cardiac disorders) | 5 | 0 | 2
CARDIAC FAILURE (Cardiac disorders) | 2 | 0 | 0
CARDIAC TAMPONADE (Cardiac disorders) | 0 | 0 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 4 | 0 | 1
SICK SINUS SYNDROME (Cardiac disorders) | 0 | 0 | 1
AORTIC VALVE DISEASE (Cardiac disorders) | 1 | 0 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 1
MITRAL VALVE STENOSIS (Cardiac disorders) | 1 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 14 | 0 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 6 | 0 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 2 | 0 | 0
HEART VALVE INCOMPETENCE (Cardiac disorders) | 0 | 0 | 1
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 1 | 0 | 0
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 | 0 | 0
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 1 | 0 | 0
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 7 | 2 | 2
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 0 | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 7 | 0 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 0 | 0
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 | 1 | 0
HYPOTENSION (Vascular disorders) | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 4 | 1 | 2
AORTIC ANEURYSM (Vascular disorders) | 1 | 0 | 0
AORTIC STENOSIS (Vascular disorders) | 1 | 0 | 0
ARTERIOSCLEROSIS (Vascular disorders) | 2 | 1 | 0
AORTIC DISSECTION (Vascular disorders) | 0 | 0 | 1
ARTERIAL STENOSIS (Vascular disorders) | 1 | 0 | 0
VENOUS THROMBOSIS (Vascular disorders) | 1 | 0 | 0
EXTREMITY NECROSIS (Vascular disorders) | 1 | 0 | 0
VASCULAR OCCLUSION (Vascular disorders) | 1 | 0 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 2 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 4 | 3 | 1
ILIAC ARTERY EMBOLISM (Vascular disorders) | 1 | 0 | 0
RHEUMATOID VASCULITIS (Vascular disorders) | 0 | 1 | 0
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 | 0 | 0
AXILLARY VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 1 | 0 | 0
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 | 0 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0 | 0
HYPERTHYROIDISM (Endocrine disorders) | 1 | 0 | 0
VICTIM OF HOMICIDE (Social circumstances) | 1 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 2 | 0 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 1 | 0
BIPOLAR DISORDER (Psychiatric disorders) | 1 | 0 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 1 | 0 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 0 | 0
HEPATITIS (Hepatobiliary disorders) | 1 | 0 | 0
CHOLANGITIS (Hepatobiliary disorders) | 1 | 0 | 0
HEPATIC MASS (Hepatobiliary disorders) | 1 | 0 | 0
LIVER INJURY (Hepatobiliary disorders) | 1 | 0 | 0
BILIARY COLIC (Hepatobiliary disorders) | 1 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 9 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 10 | 3 | 3
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 4 | 0 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 4 | 2 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 1
MIGRAINE (Nervous system disorders) | 1 | 0 | 1
SCIATICA (Nervous system disorders) | 5 | 0 | 0
NEURALGIA (Nervous system disorders) | 2 | 0 | 0
PRESYNCOPE (Nervous system disorders) | 1 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 1 | 0
RADICULOPATHY (Nervous system disorders) | 0 | 0 | 1
ENCEPHALOPATHY (Nervous system disorders) | 1 | 0 | 0
POLYNEUROPATHY (Nervous system disorders) | 1 | 0 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0 | 0
MOYAMOYA DISEASE (Nervous system disorders) | 1 | 0 | 0
NERVE COMPRESSION (Nervous system disorders) | 1 | 0 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 0 | 0
CERVICAL MYELOPATHY (Nervous system disorders) | 1 | 0 | 0
SPINAL CLAUDICATION (Nervous system disorders) | 1 | 0 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 0
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 0 | 1
NERVE ROOT COMPRESSION (Nervous system disorders) | 1 | 0 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 3 | 1 | 1
CEREBROVASCULAR DISORDER (Nervous system disorders) | 1 | 0 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 0
RUPTURED CEREBRAL ANEURYSM (Nervous system disorders) | 1 | 0 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 4 | 2 | 1
COMPLEX REGIONAL PAIN SYNDROME (Nervous system disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 1 | 0
COLITIS (Gastrointestinal disorders) | 1 | 0 | 1
VOMITING (Gastrointestinal disorders) | 2 | 2 | 0
DIARRHOEA (Gastrointestinal disorders) | 3 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 4 | 0 | 0
FAECALOMA (Gastrointestinal disorders) | 1 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 2 | 0 | 0
GINGIVITIS (Gastrointestinal disorders) | 1 | 0 | 0
ANAL FISSURE (Gastrointestinal disorders) | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 1
DIVERTICULUM (Gastrointestinal disorders) | 1 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 2 | 1 | 0
COLONIC ATONY (Gastrointestinal disorders) | 0 | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 2 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 | 2 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 5 | 0 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 2 | 1 | 0
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 | 0 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 | 1 | 0
OESOPHAGEAL SPASM (Gastrointestinal disorders) | 0 | 1 | 0
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 | 0 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 0 | 0
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 1 | 0
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 | 0 | 0
MESENTERIC ARTERY EMBOLISM (Gastrointestinal disorders) | 1 | 0 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0
ABDOMINAL HERNIA OBSTRUCTIVE (Gastrointestinal disorders) | 1 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0 | 3
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 0 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0 | 0
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 1 | 0 | 0
DEAFNESS NEUROSENSORY (Ear and labyrinth disorders) | 1 | 0 | 0
NEUROSENSORY HYPOACUSIS (Ear and labyrinth disorders) | 0 | 1 | 0
SEPSIS (Infections and infestations) | 2 | 0 | 0
ABSCESS (Infections and infestations) | 1 | 0 | 0
EMPYEMA (Infections and infestations) | 0 | 1 | 0
INFLUENZA (Infections and infestations) | 1 | 1 | 0
PNEUMONIA (Infections and infestations) | 12 | 4 | 3
SINUSITIS (Infections and infestations) | 2 | 1 | 0
UROSEPSIS (Infections and infestations) | 3 | 1 | 0
BRONCHITIS (Infections and infestations) | 10 | 3 | 0
CELLULITIS (Infections and infestations) | 6 | 1 | 1
CERVICITIS (Infections and infestations) | 1 | 0 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0 | 0
BACTERAEMIA (Infections and infestations) | 0 | 1 | 0
CANDIDIASIS (Infections and infestations) | 0 | 0 | 1
HEPATITIS E (Infections and infestations) | 0 | 1 | 0
ABSCESS LIMB (Infections and infestations) | 4 | 0 | 0
APPENDICITIS (Infections and infestations) | 5 | 0 | 0
BONE ABSCESS (Infections and infestations) | 1 | 0 | 0
EPIGLOTTITIS (Infections and infestations) | 1 | 0 | 0
OTITIS MEDIA (Infections and infestations) | 1 | 0 | 0
SEPTIC SHOCK (Infections and infestations) | 4 | 0 | 0
ASPERGILLOSIS (Infections and infestations) | 1 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 2 | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 2 | 0 | 0
TOOTH ABSCESS (Infections and infestations) | 0 | 1 | 0
BRONCHIECTASIS (Infections and infestations) | 1 | 1 | 0
DIVERTICULITIS (Infections and infestations) | 6 | 0 | 0
HERPES SIMPLEX (Infections and infestations) | 1 | 0 | 0
LUNG INFECTION (Infections and infestations) | 1 | 0 | 0
PYELONEPHRITIS (Infections and infestations) | 2 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 6 | 0 | 0
LOBAR PNEUMONIA (Infections and infestations) | 4 | 0 | 0
VIRAL INFECTION (Infections and infestations) | 1 | 0 | 0
WOUND INFECTION (Infections and infestations) | 2 | 0 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 2 | 0 | 0
SYSTEMIC MYCOSIS (Infections and infestations) | 1 | 0 | 0
BONE TUBERCULOSIS (Infections and infestations) | 1 | 0 | 0
CANDIDA PNEUMONIA (Infections and infestations) | 1 | 0 | 0
CHRONIC SINUSITIS (Infections and infestations) | 2 | 0 | 0
BURSITIS INFECTIVE (Infections and infestations) | 0 | 1 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 1 | 0 | 0
HUMAN EHRLICHIOSIS (Infections and infestations) | 1 | 0 | 0
PERIRECTAL ABSCESS (Infections and infestations) | 1 | 0 | 0
ARTHRITIS BACTERIAL (Infections and infestations) | 1 | 0 | 0
BACTERIAL INFECTION (Infections and infestations) | 0 | 0 | 1
HAEMATOMA INFECTION (Infections and infestations) | 1 | 0 | 0
INFECTED SKIN ULCER (Infections and infestations) | 0 | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 1 | 0
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 | 0 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 6 | 2 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 | 2 | 0
OSTEOMYELITIS CHRONIC (Infections and infestations) | 1 | 0 | 0
PERITONSILLAR ABSCESS (Infections and infestations) | 1 | 0 | 0
PNEUMONIA HAEMOPHILUS (Infections and infestations) | 0 | 1 | 0
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 2 | 0 | 0
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 | 0 | 0
RESPIRATORY MONILIASIS (Infections and infestations) | 1 | 0 | 0
LYMPH NODE TUBERCULOSIS (Infections and infestations) | 1 | 0 | 0
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 2 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 6 | 2 | 1
DEVICE RELATED INFECTION (Infections and infestations) | 2 | 0 | 0
INCISION SITE CELLULITIS (Infections and infestations) | 1 | 0 | 0
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 0 | 1 | 0
POST PROCEDURAL INFECTION (Infections and infestations) | 1 | 0 | 0
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 0 | 0
GASTROENTERITIS SALMONELLA (Infections and infestations) | 1 | 0 | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 1 | 0
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 0 | 0
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 0 | 0 | 1
STAPHYLOCOCCAL OSTEOMYELITIS (Infections and infestations) | 1 | 0 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 | 0 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 5 | 0 | 0
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 1 | 0 | 0
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 0 | 0 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
RENAL INFARCT (Renal and urinary disorders) | 1 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 0 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 1 | 0
RENAL AMYLOIDOSIS (Renal and urinary disorders) | 1 | 0 | 0
GLOMERULONEPHRITIS (Renal and urinary disorders) | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 5 | 0 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 3 | 0 | 0
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0 | 0
OBESITY (Metabolism and nutrition disorders) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 1 | 0
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 3 | 2 | 2
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 | 0 | 0
LYMPHADENITIS (Blood and lymphatic system disorders) | 1 | 0 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 0 | 0
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 0 | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0
BONE MARROW TOXICITY (Blood and lymphatic system disorders) | 0 | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
PANNICULITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
LICHENOID KERATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PYODERMA GANGRENOSUM (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
DERMATITIS PSORIASIFORM (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
CYSTOCELE (Reproductive system and breast disorders) | 3 | 0 | 0
ADENOMYOSIS (Reproductive system and breast disorders) | 1 | 0 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 1 | 0 | 1
OVARIAN CYST (Reproductive system and breast disorders) | 1 | 1 | 0
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 | 0 | 0
GYNAECOMASTIA (Reproductive system and breast disorders) | 0 | 1 | 0
CERVICAL POLYP (Reproductive system and breast disorders) | 1 | 0 | 0
BREAST DISORDER (Reproductive system and breast disorders) | 1 | 0 | 0
MENOMETRORRHAGIA (Reproductive system and breast disorders) | 1 | 0 | 0
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1 | 0 | 0
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0 | 0
FIBROCYSTIC BREAST DISEASE (Reproductive system and breast disorders) | 1 | 0 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 0 | 0
CONGENITAL CEREBRAL CYST (Congenital, familial and genetic disorders) | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 4 | 2 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 3 | 0 | 0
POISONING (Injury, poisoning and procedural complications) | 0 | 1 | 0
UNDERDOSE (Injury, poisoning and procedural complications) | 1 | 0 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 8 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 2 | 1 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 | 1 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
DEVICE FAILURE (Injury, poisoning and procedural complications) | 3 | 1 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 0
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 0 | 0
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 | 0 | 0
STRESS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
MEDICATION ERROR (Injury, poisoning and procedural complications) | 1 | 0 | 0
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 2 | 0 | 0
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 2 | 1 | 1
BURNS THIRD DEGREE (Injury, poisoning and procedural complications) | 0 | 1 | 0
DEVICE DISLOCATION (Injury, poisoning and procedural complications) | 1 | 0 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 3 | 1 | 0
PUBIC RAMI FRACTURE (Injury, poisoning and procedural complications) | 1 | 2 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
LIMB CRUSHING INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
TRAUMATIC LIVER INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
DISLOCATION OF VERTEBRA (Injury, poisoning and procedural complications) | 1 | 0 | 0
DRUG ADMINISTRATION ERROR (Injury, poisoning and procedural complications) | 1 | 0 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 1 | 0
THERAPEUTIC AGENT TOXICITY (Injury, poisoning and procedural complications) | 1 | 0 | 0
INCORRECT DOSE ADMINISTERED (Injury, poisoning and procedural complications) | 2 | 0 | 0
MEDICAL DEVICE COMPLICATION (Injury, poisoning and procedural complications) | 1 | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 2 | 2 | 0
SUTURE RELATED COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0 | 0
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 2 | 0 | 0
DISLOCATION OF JOINT PROSTHESIS (Injury, poisoning and procedural complications) | 2 | 0 | 0
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 10 | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 | 1 | 2
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
BONE EROSION (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 8 | 0 | 0
HAND DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 27 | 3 | 2
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
JOINT ANKYLOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
FINGER DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
JOINT DESTRUCTION (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
RHEUMATOID NODULE (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 56 | 21 | 9
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 7 | 2 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
BRONCHIAL POLYP (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RHEUMATOID LUNG (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
TRACHEAL STENOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
STATUS ASTHMATICUS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
DEATH (General disorders) | 1 | 1 | 0
HERNIA (General disorders) | 1 | 0 | 0
FATIGUE (General disorders) | 1 | 0 | 0
MALAISE (General disorders) | 1 | 0 | 0
PYREXIA (General disorders) | 4 | 1 | 1
ASTHENIA (General disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 13 | 4 | 3
HYPERTHERMIA (General disorders) | 1 | 1 | 0
IMPAIRED HEALING (General disorders) | 1 | 0 | 0
HERNIA OBSTRUCTIVE (General disorders) | 1 | 0 | 0
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
OSTEOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1 | 2
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
ADENOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
LEIOMYOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
KAPOSI'S SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
SEBACEOUS CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 5 | 3
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
BREAST CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 1 | 0
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
CERVIX CARCINOMA STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 2 | 0
SQUAMOUS CELL CARCINOMA OF THE CERVIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
SMALL CELL LUNG CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
EXTRANODAL MARGINAL ZONE B-CELL LYMPHOMA (MALT TYPE) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label (OL) Abatacept (N=1184) | Abatacept (ABA) (N=959) | Placebo (PLA) (N=482)
CONJUNCTIVITIS (Eye disorders) | 72 | 22 | 11
HYPERTENSION (Vascular disorders) | 162 | 68 | 24
INSOMNIA (Psychiatric disorders) | 96 | 43 | 14
DEPRESSION (Psychiatric disorders) | 76 | 37 | 13
HEADACHE (Nervous system disorders) | 216 | 195 | 69
DIZZINESS (Nervous system disorders) | 135 | 105 | 43
NAUSEA (Gastrointestinal disorders) | 154 | 121 | 56
VOMITING (Gastrointestinal disorders) | 101 | 58 | 27
DIARRHOEA (Gastrointestinal disorders) | 186 | 96 | 58
DYSPEPSIA (Gastrointestinal disorders) | 112 | 72 | 24
ABDOMINAL PAIN (Gastrointestinal disorders) | 96 | 35 | 16
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 101 | 44 | 18
RHINITIS (Infections and infestations) | 67 | 28 | 7
INFLUENZA (Infections and infestations) | 145 | 60 | 30
SINUSITIS (Infections and infestations) | 198 | 66 | 35
BRONCHITIS (Infections and infestations) | 229 | 52 | 25
PHARYNGITIS (Infections and infestations) | 90 | 22 | 12
GASTROENTERITIS (Infections and infestations) | 87 | 14 | 7
NASOPHARYNGITIS (Infections and infestations) | 266 | 98 | 46
URINARY TRACT INFECTION (Infections and infestations) | 195 | 78 | 23
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 362 | 143 | 74
ANAEMIA (Blood and lymphatic system disorders) | 65 | 18 | 14
RASH (Skin and subcutaneous tissue disorders) | 85 | 45 | 19
MYALGIA (Musculoskeletal and connective tissue disorders) | 69 | 33 | 19
BACK PAIN (Musculoskeletal and connective tissue disorders) | 210 | 68 | 28
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 70 | 21 | 13
COUGH (Respiratory, thoracic and mediastinal disorders) | 195 | 84 | 37
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 77 | 18 | 5
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 80 | 30 | 25
FATIGUE (General disorders) | 63 | 65 | 25
PYREXIA (General disorders) | 65 | 37 | 18
CHEST PAIN (General disorders) | 73 | 26 | 11
OEDEMA PERIPHERAL (General disorders) | 83 | 35 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.